CLINICAL TRIAL: NCT02230332
Title: Proof of Concept Study of Alendronate for Asthma
Brief Title: Alendronate to Prevent Loss of Bronchoprotection in Asthma
Acronym: ALFA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, dave mauger, Professor of Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AsthmaNet 009; U10HL098115 (NIH)
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Results first posted 2017-12-14 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2017-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Alendronate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alendronate (Experimental): Alendronate in 10mg capsules taken once daily
  Interventions: Drug: Alendronate
- Placebo (Placebo Comparator): Placebo capsule taken once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alendronate
  Other Names: Fasomax
  Arms: Alendronate
Drug: Placebo
  Arms: Placebo

SUMMARY:
Beta-2-agonists are effective in reducing airway narrowing in asthma and protecting against stimuli that produce bronchoconstriction. The combination of long-acting beta agonists (LABA) and inhaled corticosteroids (ICS) has become the most commonly used asthma controller medication class in the United States, but unfortunately, even when LABAs are added to ICS and used regularly, 58-81% of patients with asthma fail to achieve total control. Regular use of beta-agonists, both short and long-acting, reduces the ability of these agents to protect against the airway narrowing that occurs in asthma in response to bronchoconstrictor stimuli. We refer to this reduced effect as loss of bronchoprotection. In this proof of concept trial we aim to determine if alendronate, which diminishes beta-2 adrenergic receptor internalization, can reduce the loss of bronchoprotection that occurs with regular use of LABAs, even when used in combination with ICS.

ELIGIBILITY:
Inclusion Criteria:

* Clinical history consistent with moderate asthma for >1 year
* Asthma is controlled with ICS, with an FP dose ≤ 1000mcg/day and >100mcg/day (or equivalent)
* Able to perform reproducible spirometry according to ATS criteria
* Baseline FEV1 ≥ 50% of predicted and ≥1L.
* If FEV1 <80%, a minimum 12% increase in FEV1 post-bronchodilator or a MCh PC20 ≤ 8 mg/mL
* If FEV1 ≥80%, a MCh PC20 ≤ 8 mg/mL
* Salmeterol protected MCh ≤ 16 mg/mL

Exclusion Criteria:

* Uncontrolled asthma, as suggested by an ACT score <18 while on high-dose ICS (FP daily dose >500mcg or equivalent)
* Non-ICS controller medication or LABA use within 4 weeks of study entry.
* Contraindications to use of bisphosphonates: history of intolerance to bisphosphonates, history of esophageal ulcers, history of hematemesis, uncontrolled gastro-esophageal reflux disease, inability to stay erect for 30 minutes after oral drug, history of osteonecrosis of the jaw, dental extraction or root canal in prior 8 weeks, or anticipated during the study
* Calculated GFR of less than 35 mL/min
* History of smoking (cigarettes, cigars, pipes, marijuana or any other substances) within the past 1 year, or > 10 pack-years total if ≥ 18 years of age
* Systemic corticosteroid treatment for any condition within 4 weeks of enrollment at Visit 1, history of significant asthma exacerbation requiring systemic corticosteroids within 4 weeks of Visit 1 or more than five courses of systemic corticosteroids in the past year, history of a life-threatening asthma exacerbation requiring intubation, mechanical ventilation, or resulting in a hypoxic seizure within the last 2 years
* History of a respiratory tract infection within 4 weeks of Visit 1
* Receiving hyposensitization therapy other than an established maintenance regimen defined as a continuous regimen for ≥ 3 months prior to enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos Cardet, MD, Study Director — Brigham and Women's Hospital
Locations (10):
- United States (10):
  - University of Arizona College of Medicine, Tucson, Arizona
  - University of California - San Francisco, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Cardet JC, Jiang X, Lu Q, Gerard N, McIntire K, Boushey HA, Castro M, Chinchilli VM, Codispoti CD, Dyer AM, Holguin F, Kraft M, Lazarus S, Lemanske RF, Lugogo N, Mauger D, Moore WC, Moy J, Ortega VE, Peters SP, Smith LJ, Solway J, Sorkness CA, Sumino K, Wechsler ME, Wenzel S, Israel E; AsthmaNet Investigators. Loss of bronchoprotection with ICS plus LABA treatment, beta-receptor dynamics, and the effect of alendronate. J Allergy Clin Immunol. 2019 Aug;144(2):416-425.e7. doi: 10.1016/j.jaci.2019.01.049. Epub 2019 Mar 11. PMID 30872116
- See also: AsthmaNet home page — http://asthmanetresearch.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were recruited from the community between January 2015 and May 2016 at 9 U.S. sites from the NHLBI AsthmaNet research network.
Pre-assignment Details: Participants with persistent asthma were first treated with fluticasone propionate 250mcg twice daily for 2 weeks during the run-in. Most of the participants who were not randomized did not meet the Salmeterol Protected Methacholine Challenge inclusion criterion.
Groups:
- Alendronate: Alendronate in 10mg capsules taken once daily
  Alendronate
- Placebo: Placebo capsule taken once daily
  Placebo
Period: Overall Study
Arm/Group | Alendronate | Placebo
Started | 38 | 40
Completed | 34 | 39
Not Completed | 4 | 1
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alendronate | Placebo | Total
Number analyzed (Participants) | 38 | 40 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (13.1) | 39.3 (12.3) | 38.8 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 27 | 47
  Male | 18 | 13 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 24 | 21 | 45
  Black | 10 | 13 | 23
  Asian/Pacific Islander | 1 | 3 | 4
  Hispanic or Latio | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 38 | 40 | 78
Asthma Control Test score [Mean (Inter-Quartile Range); unit: units on a scale] — Asthma Control Test : Score calculated as the sum total of a 5-item questionnaire. Each item ranges from 1 (poor control) to 5 (good control) so that the range of the total score is 5 to 25. Scores below 20 indicate that asthma is not well controlled.
  units on a scale | 21 [18 to 23] | 21 [19 to 23] | 21 [19 to 23]
FEV1 - percent of predicted [Mean (Standard Deviation); unit: percent of predicted] | 81.3 (14.9) | 83.1 (14.0) | 82.2 (14.4)
Salmeterol Protected Methcholine PC20 [Geometric Mean (Standard Deviation); unit: mg/ml] — During the challenge, the patient inhales methacholine aerosols in increasing concentrations. Spirometry is performed before and after each methacholine dose, and the results are reported as a percent decrease in FEV1 from baseline for each increasing dose of methacholine. A positive reaction to methacholine is a 20% fall in FEV1, and the provocative concentration that causes a positive reaction (the PC20) is used to indicate the level of airway hyperresponsiveness. Smaller numbers indicate greater airway hyperresponsiveness.
  mg/ml | 5.4 (0.8) | 3.7 (1) | 4.5 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Salmeterol Protected Methacholine Challenge PC20
Description: Following administration of Salmeterol, the concentration of Methacholine required to produce a 20% drop in FEV1 - measured in mg/ml and reported on log base 2 scale.
Time Frame: 8 weeks after randomization
Measure: Mean (95% Confidence Interval); unit: mg/ml on log base 2 scale
Arm/Group | Alendronate | Placebo
Number analyzed (Participants) | 34 | 39
mg/ml on log base 2 scale | 1.8 [1.1 to 2.5] | 1.7 [1.1 to 2.3]

2. Secondary Outcome: Peripheral Blood Mononuclear Cell ADRB2 Cell Surface Density
Time Frame: 8 weeks after randomization
Measure: Geometric Mean (95% Confidence Interval); unit: number of receptors per cell
Arm/Group | Alendronate | Placebo
Number analyzed (Participants) | 34 | 39
number of receptors per cell | 1680 [1359 to 2076] | 1863 [1473 to 2358]

3. Secondary Outcome: Beta-2 Adrenergic Receptor Agonist-induced cAMP Production
Description: Peripheral blood mononuclear cells cAMP concentrations measured using isoproterenol (ISO) as a beta-2 adrenergic receptor agonist, and using phosphate buffered saline (PBS) as a positive control. The outcome is expressed as the ratio of cAMP concentration using ISO relative to cAMP concentration using PBS.
Time Frame: 8 weeks after randomization
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Alendronate | Placebo
Number analyzed (Participants) | 34 | 39
ratio | 5.9 [4.7 to 7.5] | 5.9 [4.9 to 7.2]

4. Other Pre Specified Outcome: Salivary Alpha Amylase Ratio (Post-Salmeterol / Pre-Salmeterol)
Description: Salivary Alpha Amylase (sAA) levels from saliva samples obtained through passive drooling, before and 1 hour after Salmeterol administration. The outcome is expressed as the ratio of the Post-Salmeterol to the Pre-Salmeterol sAA levels.
Time Frame: 8 weeks after randomization
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Alendronate | Placebo
Number analyzed (Participants) | 34 | 39
ratio | 1.6 [1.4 to 1.9] | 1.6 [1.3 to 1.9]

5. Other Pre Specified Outcome: Asthma Control Test (ACT)
Description: Asthma Control Test : Score calculated as the sum total of a 5-item questionnaire. Each item ranges from 1 (poor control) to 5 (good control) so that the range of the total score is 5 to 25. Scores below 20 indicate that asthma is not well controlled.
Time Frame: 8 weeks after randomization
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Alendronate | Placebo
Number analyzed (Participants) | 34 | 39
units on a scale | 22.2 [21.2 to 23.2] | 22.2 [21.4 to 23.1]

6. Other Pre Specified Outcome: Fractional Exhaled Nitrix Oxide
Time Frame: 8 weeks after randomization
Measure: Geometric Mean (95% Confidence Interval); unit: parts per billion
Arm/Group | Alendronate | Placebo
Number analyzed (Participants) | 34 | 39
parts per billion | 16.8 [12.9 to 21.9] | 15.4 [11.7 to 20.1]

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Alendronate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/38 | 2/40
Other Adverse Events (participants affected / at risk) | 9/38 | 13/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alendronate (N=38) | Placebo (N=40)
Viral Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
GI Bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alendronate (N=38) | Placebo (N=40)
Esophageal reflux (Gastrointestinal disorders) | 2 (2) | 0 (0)
Acute nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Acute sinusitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Acue Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
thrush (Infections and infestations) | 0 (0) | 2 (2)
headache (General disorders) | 2 (2) | 4 (5)
Heartburn (General disorders) | 2 (2) | 0 (0)
Nausea alone (General disorders) | 0 (0) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No